CLINICAL TRIAL: NCT05114057
Title: Use of NGAL to Optimize Fluid Dosing, CRRT Initiation and Discontinuation in Critically Ill Children and Neonates with Acute Kidney Injury
Brief Title: Use of NGAL for Fluid Dosing and CRRT Initiation in Pediatric and Neonatal AKI
Acronym: Taking Focus 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CIN002 - Taking Focus 3
Record Dates: First submitted 2021-10-20; First posted 2021-11-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury; Acute Kidney Injury Due to Sepsis; Neonatal Sepsis
Keywords: Renal Angina Index; NGAL
MeSH Terms: conditions — Acute Kidney Injury; Neonatal Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PICU Patients (Other): Prospectively enrolled patients admitted to the PICU will be assessed by the RAI calibration for sepsis in the PICU and including additional risk factors.
  Interventions: Other: Renal Angina Index (RAI)
- CICU Patients (Other): Prospectively enrolled patients admitted to the CICU will be assessed by the RAI calibration specific to the CICU, especially post cardiac bypass
  Interventions: Other: Renal Angina Index (RAI)
- NICU Patients (Other): Prospectively enrolled patients admitted to the NICU will be assessed by the RAI calibration for neonatal patients with sepsis or post abdominal surgeries
  Interventions: Other: Renal Angina Index (RAI)

INTERVENTIONS:
Other: Renal Angina Index (RAI) — Risk-stratification tool using measures of risk and presence of injury to predict Acute Kidney Injury

SUMMARY:
This study will follow patients admitted to the PICU with sepsis, NICU with sepsis or after abdominal surgery, or CICU who are identified as being at risk for developing acute kidney injury. The investigators will use risk-stratification, biomarker testing, and a functional assessment to predict children and neonates who will become fluid overloaded and develop severe acute kidney injury.

DETAILED DESCRIPTION:
In the pediatric population, acute kidney injury (AKI) is commonly observed in critically ill patients. At this time, there are no standardized care pathways that begin at identifying patients at risk for developing AKI and progress through to early recognition and treatment. Through previous work, the investigators have integrated a risk-stratification tool (renal angina index or RAI) and a urine biomarker (NGAL) to try to identify PICU patients at risk versus not at-risk for developing AKI. Through this study, the investigators will tailor the RAI to the septic population in the PICU, create a new NICU RAI, and investigate the utility of the CICU specific RAI in a prospective population. Biomarker testing will be used to further risk-stratify those patients deemed at highest risk through the RAI.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Pediatric Intensive Care Unit (PICU), Cardiac Intensive Care Unit (CICU), or Neonatal Intensive Care Unit (NICU) at participating institution

Exclusion Criteria:

* Baseline Chronic Kidney Disease (CKD) Stage IV or V (estimated GFR <60 mL/min/1.736m2)
* History of kidney transplant within the previous 90 days
* Ongoing AKI or Acute Kidney Disease (AKD) at ICU admission requiring renal replacement therapy initiated prior to ICU admission
* Acute DNR order or clinical team is not committed to escalating medical care
* Anticipated to require intensive care for less than 48 hours

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1380 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Decision Support Performance | Days 2-4 after ICU admission
  Accuracy of the risk stratification and biomarker testing to rule out Acute Kidney Injury at ICU Days 2-4 as measured by the negative predictive value (NPV)

SECONDARY OUTCOMES:
Rate of Clinical Decision Support Completion | 48 hours
  Time to complete the risk stratification and biomarker testing is less than 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stuart L Goldstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided